CLINICAL TRIAL: NCT02193126
Title: Permanency Innovations Initiative- Trauma Focus Model for Reducing Long-Term Foster Care Project
Brief Title: Trauma Focus Model for Reducing Long-Term Foster Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Westat (Other)
Collaborators: Children's Bureau - Administration for Children and Families (Other); Illinois Department of Children and Family Services. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Other
Other Study IDs: 8977 3
Record Dates: First submitted 2014-07-09; First posted 2014-07-17 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Foster Care
Keywords: Long term foster care; child abuse and neglect; trauma
MeSH Terms: conditions — Wounds and Injuries | interventions — Educational Status; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Other: Trauma Affect Regulation: Guide for Education and Therapy (TARGET)
- Comparison (No Intervention)

INTERVENTIONS:
Other: Trauma Affect Regulation: Guide for Education and Therapy (TARGET) — The intervention is called the Trauma Affect Regulation: Guide for Education and Therapy (TARGET). TARGET is a manualized, psycho-educational intervention delivered in 10 - 12 sessions. TARGET is designed to address complex trauma and difficulties with emotional regulation and relational engagement that occur across a wide range of trauma-related difficulties, including trauma-related and behavioral symptoms. The full TARGET model consists of learning 7 essential core skills. These skills are called the FREEDOM steps: Focus, Recognize triggers, Emotion self-check, Evaluate thoughts, Define goals, Options, and Make a contribution.
  Other Names: TARGET
  Arms: Treatment

SUMMARY:
The Trauma Focus Model for Reducing Long-Term Foster Care Project with the Illinois Department of Children and Family Services (DCFS) is implementing a trauma-focused intervention, Trauma Affect Regulation: Guide for Education and Therapy (TARGET) to increase permanency rates for a target population of children identified as being most at risk of long-term foster care.

DETAILED DESCRIPTION:
The Illinois Department of Children and Family Services (DCFS) is one of six recipients of the Permanency Innovations Initiative Grant. These funds support the statewide implementation of Trauma Affect Regulation: Guide for Education and Therapy (TARGET) in Illinois. TARGET is a manualized, psycho-educational intervention designed to address complex trauma and difficulties with emotional regulation and relational engagement that occur across a wide range of trauma-related difficulties, including trauma-related and behavioral symptoms. The aim of this intervention is to address the key barriers to permanence for the target population. This population includes youth ages 11-16 who are placed in traditional, relative, and specialized foster homes throughout the state of Illinois, have been in foster care for at least 2 years, and are experiencing mental health challenges and/or at least one placement change. The three key barriers to permanency are: (1) children's need to improve emotional regulation and reduce symptom severity, particularly disruptive behaviors; (2) biological parents' skills in regulating their emotions so they are better able to complete services and address the underlying issues related to their involvement in the child welfare system; (3) foster parents and other placement resources skills in understanding and addressing the needs and disruptive behaviors of the children in their care with trauma histories.

The local evaluation will examine the effectiveness of the TARGET program in increasing permanency rates for foster youth in the target population. The main hypothesis to be tested is that addressing unstable child affect & behavior secondary to trauma using an intervention that improves both youth modulation skills as well as foster parent capacity to respond appropriately to youth will stabilize placements and improve youth ability to engage with potential permanency resources, thus facilitating progress toward permanence. The evaluation involves randomly assigning eligible foster youth to receive TARGET services or receive services as usual. The evaluators collect proximal and distal outcomes from multiple administrative data sources. Additionally, the evaluation includes the collection of key proximal outcomes through the use of interviews with foster youth, their foster parents and biological parents deemed eligible for participation in the project.

ELIGIBILITY:
Inclusion Criteria:

* Youth ages 11-16 who are placed in traditional, relative, and specialized foster homes throughout the state of Illinois who, upon reaching the two-year anniversary of entering care, are experiencing mental health symptoms and/or have had at least one placement change.
* If a youth does not exhibit any mental health symptoms as indicated by the Child and Adolescent Needs and Strength (CANS) tool, they need to have at least 3 placement changes to be eligible for the study.

Exclusion Criteria:

* Youth are ineligible to participate if at the time of eligibility assessment, they are in need of immediate and acute substance abuse treatment, have a Full Scale IQ score below 70, and/or have made recent suicidal threats or plans.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 462 (Actual)
Dates: Start 2014-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Time to stable permanence | Measured from the date of random assignment to the discharge date or to the end of the study period for cases that did not discharge
  Measured by administrative data from the Adoption and Foster Care Analysis and Reporting System (AFCARS)
Placement stability | Measured at initial study enrollment and at the 8, 14, 20, and 26-month mark of enrollment in the study
  Measured by administrative data from the Adoption and Foster Care Analysis and Reporting System (AFCARS)

SECONDARY OUTCOMES:
Foster parent skills in responding to youth's emotional and behavioral dysregulation | completed by study youth at initial study enrollment and at 6 months after baseline data collection
  Measured by Parenting Practices Chicago Survey (PPCS) (Gorman-Smith et al., 1996)

OTHER OUTCOMES:
Biological parent ability to regulate their own emotions and behaviors and experience of trauma-related symptoms | completed by biological parents of study youth at initial study enrollment and at 6 months after baseline data collection
  Measured by Abbreviated Dysregulation Inventory (ADI) (Mezzich et al., 2001)
Biological parent service completion | Measured at initial study enrollment and at the 8, 14, 20, and 26-month mark of enrollment in the study
  Measured by administrative data from the Administrative Case Review (ACR)
Biological parent contact with youth | completed by study youth at initial study enrollment and at 6 months after baseline data collection
  Measured by Parent Contact with Youth (PCY) Instrument (questions modified from the Illinois Adult Connections Study)
Change in Youth trauma-related and mental health symptoms | 1) Measured at initial study enrollment and at the 8, 14, 20, and 26-month mark of enrollment in the study and 2) completed by study youth at initial study enrollment and at 6 months after baseline data collection
  Measured by: 1) administrative data from the Child and Adolescent Needs and Strength (CANS) tool and 2) the Trauma Symptoms Checklist for Children (TSCC) (Briere, 1996)
Youth capacity to form and maintain relationships. | Measured 1) at initial study enrollment and at the 8, 14, 20, and 26-month mark of enrollment in the study and 2) completed by study youth at initial study enrollment and at 6 months after baseline data collection
  Measured by: 1) administrative data from the Child and Adolescent Needs and Strength (CANS) tool and 2) Youth Social Support Instrument (YSS) (LONGSCAN, 1998)
Youth capacity to regulate their emotions and behavior | Measured 1) at initial study enrollment and at the 8, 14, 20, and 26-month mark of enrollment in the study and 2) completed by both study youth and their current caregiver at initial study enrollment and at 6 months after baseline data collection
  Measured by: 1) administrative data from the Child and Adolescent Needs and Strength (CANS) tool and 2) the Abbreviated Dysregulation Inventory (ADI) (Mezzich et al., 2001)
Change in support for biological and foster parents | Measured at initial study enrollment and at 6 months after baseline data collection
  Measured by Social Provisions Scale (SPS) (Russell & Cutrona, 1984) completed by both biological and foster parents of study youth
Change in Youth traumatic events | Measured at initial study enrollment and at the 8, 14, 20, and 26-month mark of enrollment in the study
  Measured by administrative data from the Child and Adolescent Needs and Strength (CANS) tool
Youth emotional permanency | Measured at initial study enrollment and at 6 months after baseline data collection
  Measured by Youth Emotional Permanency (YEP) Instrument (questions from the current Illinois Adult Connections Study and the Supportive Connections Inventory developed for the Arizona PII evaluation) completed by youth
Frequencies of change in direction of youth permanency | collected at 6, 12, 18, and 24 months
  Measured by administrative data from the Integrated Database (IDB)
Permanency rates | collected at 6, 12, 18, and 24 months
  Measured by administrative data from the Adoption and Foster Care Analysis and Reporting System (AFCARS) collected every 6 months throughout the study duration.
Timely permanence | collected at 6, 12, 18, and 24 months
  Measured by administrative data from the Adoption and Foster Care Analysis and Reporting System (AFCARS)
Placement stability after legal permanency | collected at 6, 12, 18, and 24 months
  Measured by administrative data from the Adoption and Foster Care Analysis and Reporting System (AFCARS)
Repeat maltreatment following legal permanence | collected at 6, 12, 18, and 24 months
  Measured by administrative data from the Adoption and Foster Care Analysis and Reporting System (AFCARS)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Sedlak, PhD., Study Director — Westat; Mark Testa, PhD., Principal Investigator — University of North Carolina